CLINICAL TRIAL: NCT02902666
Title: A Single Dose Bioequivalence Study of Test Product (One Tablet of Paracetamol 1000 mg + Codeine 30 mg, Manufactured by A.C.R.A.F. S.p.A.) vs. Two Tablets of the Reference Product (Paracetamol 500 mg + Codeine 30 mg) in Healthy Volunteers
Brief Title: Bioequivalence Study of One Tablet of Paracetamol 1000 mg + Codeine 30 mg vs. Two Tablets of Paracetamol 500 mg + Codeine 30 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 044(1F)PO15313; CRO-PK-15-304 (Other: CROSS Research S.A., Phase I Unit)
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Paracetamol 1000 mg/codeine 30 mg; Co-efferalgan 500 mg/30 mg
MeSH Terms: interventions — Acetaminophen; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol 1000 mg/codeine phosphate hemihydrate 30 mg tablet (Experimental): A single dose of the experimental drug will be administered to healthy male and female volunteers under fasting conditions before (treatment arm 1) or after (treatment arm 2) a wash-out interval of at least 7 days between the active comparator administration.
  Test formulation will be administered as a single dose of one paracetamol 1000 mg/codeine 30 mg tablet.
  Interventions: Drug: Paracetamol 1000 mg/codeine phosphate hemihydrate 30 mg tablet
- paracetamol 500mg/codeine phosphate hemihydrate 30mg 2 tablets (Active Comparator): A single dose of active comparator will be administered to healthy male and female volunteers under fasting conditions before (treatment arm 2) or after (treatment arm 1) a wash-out interval of at least 7 days between the experimental drug administration. Reference formulation will be administered as a single dose of two 500 mg/30 mg tablets.
  Interventions: Drug: Paracetamol 500 mg/codeine phosphate hemihydrate 30 mg tablet

INTERVENTIONS:
Drug: Paracetamol 1000 mg/codeine phosphate hemihydrate 30 mg tablet
  Arms: Paracetamol 1000 mg/codeine phosphate hemihydrate 30 mg tablet
Drug: Paracetamol 500 mg/codeine phosphate hemihydrate 30 mg tablet
  Arms: paracetamol 500mg/codeine phosphate hemihydrate 30mg 2 tablets

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a new paracetamol 1000 mg/codeine 30 mg formulation vs. the marketed reference Co-efferalgan® 500 mg/30 mg in terms of rate and extent of absorption, when administered as single oral dose (one tablet of the new A.C.R.A.F. formulation vs. two tablets of the reference formulation Co-efferalgan®) to healthy male and female volunteers, under fasting conditions, in two consecutive study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females, 18-55 years old inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Tobacco: non-smokers or ex-smokers for at least 6 months
7. Contraception and fertility (females only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner. Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening.

Exclusion Criteria:

1. Electrocardiogram (12-leads, supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle (paracetamol and/or codeine) and/or formulations' ingredients or related drugs, namely non-steroidal anti-inflammatory agents and/or opioid derivatives; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, genitourinary, cardiovascular, respiratory (including allergic asthma, allergic or chronic bronchitis and other pulmonary diseases), skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) medications and herbal remedies for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2010], caffeine (>5 cups coffee/tea/day) abuse
10. Drug test: positive result at the drug test at screening or day-1
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cmax of both paracetamol and codeine after administration of one tablet of a new paracetamol 1000 mg/codeine 30 mg formulation vs. two tablets of the marketed reference Co-efferalgan® 500 mg/30 mg (dose normalisation will be applied for codeine). | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
  Maximum plasma concentration (μg/ml)
AUC(0-t) of both paracetamol and codeine after administration of one tablet of a new paracetamol 1000 mg/codeine 30 mg formulation vs. two tablets of the marketed reference Co-efferalgan® 500 mg/30 mg (dose normalisation will be applied for codeine). | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
  Area under the plasma concentration-time curve from administration time to the time (t) of the last measurable concentration (Ct), calculated with the linear trapezoidal method (μg*h/ml)

SECONDARY OUTCOMES:
Area under the concentration vs. time curve up to infinity (AUC(0-∞)) of paracetamol and of codeine (free base) after single dose administration of T and R (dose normalisation will be applied to AUC(0-∞), for codeine) | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
Time to achieve Cmax (h) (Tmax) of paracetamol and of codeine (free base) after single dose administration of T and R (dose normalisation will be applied to AUC(0-∞), for codeine) | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
Terminal half-life, calculated, if feasible, as ln2/λz [h] (t1/2,z) of paracetamol and of codeine (free base) after single dose administration of T and R (dose normalisation will be applied to AUC(0-∞), for codeine) | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
Apparent First Order Terminal Rate Constant (λz) of paracetamol and of codeine (free base) after single dose administration of T and R (dose normalisation w | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
Time Until First Nonzero Concentration (tlag) of paracetamol and of codeine (free base) after single dose administration of T and R (dose normalisation will be applied to AUC(0-∞), for codeine) | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose
Treatment-Emergent Adverse Event (TEAEs), vital signs (BP, HR), physical examinations, laboratory parameters, body weight, ECG | 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.

IPD SHARING:
Plan to Share IPD: No